CLINICAL TRIAL: NCT00821054
Title: An Open Label Study to Examine the Effects of Low-Fat and High-Fat Meals on the Pharmacokinetics of Orally Administered Lapatinib in Metastatic ErbB2 Positive Breast Cancer Patients
Brief Title: A Study to Examine the Effects of Low and High-fat Meals on Orally Administered Lapatinib in Metastatic ErbB2 Positive Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 111582
Record Dates: First submitted 2008-12-18; First posted 2009-01-12 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms, Breast
Keywords: Phase I Food Effect
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

ARMS (3):
- Period 1 (Experimental): Treatment A, B or C
  Interventions: Drug: Lapatinib
- Period 2 (Experimental): Treatment A, B or C
  Interventions: Drug: Lapatinib
- Period 3 (Experimental): Treatment A, B or C
  Interventions: Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib — Treatment A: one dose of 1250mg lapatinib 1 hour before starting a low-fat breakfast; Treatment B: one dose of 1250mg lapatinib 1 hour after finishing a low fat breakfast; or Treatment C: one dose of 1250mg lapatinib 1 hour after finishing a high-fat breakfast.
  Other Names: TYKERB - US; TYVERB - UK

SUMMARY:
This study will be a randomized 3-treatment, cross-over study to evaluate the bioavailability of lapatinib administered after a high or low-fat meal.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, histologically confirmed breast cancer that over-expresses ErbB2 (3+ by IHC; FISH or CISH positive).
* Is at least 18 years of age and not greater than 65 years of age.
* Is male or female. A female is eligible to enter and participate in the study if she is of:

  1. Non-childbearing potential (i.e. physiologically incapable of becoming pregnant), including any female who: has had a hysterectomy; has had a bilateral oophorectomy (ovariectomy); has had a bilateral tubal ligation, or is post-menopausal (a demonstration of total cessation of menses for ≥ 1 year) or in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory.
  2. Childbearing potential, has a negative serum pregnancy test at Screening and agrees to one of the following: double-barrier contraception (condom with spermicidal jelly, foam, suppository, or film; diaphragm with spermicide; or male condom and diaphragm); complete abstinence from sexual intercourse from two weeks prior to administration of the study drug, throughout the active study treatment period; vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
* Is able to swallow and retain oral medication.
* ECOG performance status 0 to 2.
* Adequate bone marrow function.
* Hemoglobin ≥ 9 gm/dL.
* Absolute granulocyte count ≥1,500/mm3 (1.5 x 109/L).
* Platelets ≥ 75,000/mm3 (75 x 109/L).
* Calculated creatinine clearance (CrCl) ≥ 50 ml/min based on Cockcroft and Gault
* Total bilirubin ≤ 1.5 X upper limit of normal of institutional values and INR ≤ 1.5.
* Alanine transaminase (ALT) ≤ three times the upper limit of the institutional values or ≤ five times ULN with documented liver metastases.
* Has a left ventricular ejection fraction (LVEF) within the normal institutional range based on ECHO or MUGA.
* Life expectancy of ≥12 weeks
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Is pregnant or lactating.
* Has malabsorption syndrome, a disease affecting gastrointestinal function, or resection of the stomach or small bowel.
* Has current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
* Has evidence of symptomatic or uncontrolled brain metastases or leptomeningeal disease. Subjects with brain metastases treated by surgery and/or radiotherapy are eligible if neurologically stable and do not require steroids or anticonvulsants.
* Is considered medically unfit for the study by the investigator as a result of the medical interview, physical exam, or screening investigations.
* Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the investigational product such as gefitinib [Iressa] and erlotinib [Tarceva].
* Has received treatment with any investigational drug in the previous four weeks.
* Has received chemotherapy, immunotherapy, biologic therapy or hormonal therapy for the treatment of cancer within the past 14 days, with the exception of mitomycin C which is restricted for the past six weeks.
* Is receiving any prohibited medication within the timeframe indicated on the prohibited medication list for this study.
* Has physiological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Has inadequate venous access for protocol-related blood draws.
* Clinically significant electrocardiogram (ECG) abnormality.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Has consumed red wine, seville oranges, grapefruit or grapefruit juice and/or kumquats, pummelos, exotic citrus fruit (i.e. star fruit, bitter melon), grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-03-06 (Actual); Primary Completion 2011-03-22 (Actual); Study Completion 2011-03-22 (Actual)

PRIMARY OUTCOMES:
Protocol specified pharmacokinetic parameters | 3 weeks

SECONDARY OUTCOMES:
Safety and tolerability as assessed by evaluation of adverse events (AEs), changes in laboratory values, and vital signs | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (2):
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Greenville, South Carolina
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Amsterdam, Netherlands

REFERENCES:
- [Derived] Devriese LA, Koch KM, Mergui-Roelvink M, Matthys GM, Ma WW, Robidoux A, Stephenson JJ, Chu QS, Orford KW, Cartee L, Botbyl J, Arya N, Schellens JH. Effects of low-fat and high-fat meals on steady-state pharmacokinetics of lapatinib in patients with advanced solid tumours. Invest New Drugs. 2014 Jun;32(3):481-8. doi: 10.1007/s10637-013-0055-4. Epub 2013 Dec 19. PMID 24346280
- See also: Results for study 111582 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111582?search=study&search_terms=111582#rs